CLINICAL TRIAL: NCT01602055
Title: A Bioequivalence Study of Two Azithromycin Tablet Formulations in Indonesian Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PT Novell Pharmaceutical Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: XXI/32/CL/2009
Record Dates: First submitted 2012-05-15; First posted 2012-05-18 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Fasting
MeSH Terms: conditions — Fasting | interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azivol (Experimental)
  Interventions: Drug: Azithromycin
- Zithromax (Active Comparator)
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Single dose 500 mg of film coated tablet
  Arms: Azivol
Drug: Azithromycin — Single dose 500 mg of film coated tablet
  Arms: Zithromax

SUMMARY:
The aim of this study is to assess the bioequivalence of 500 mg Azithromycin FC tablets (Azivol) produced by PT. Novell Pharmaceutical Laboratories, compared to the reference product Zithromax 500 mg FC tablet produced by Pfizer Australia Pty, Ltd

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, both sexes, age between 18 to 55 years old
* Weight with normal range according to accepted normal values for BMI (18-25 kg/m2)
* Give a written informed consent
* Acceptable medical history and physical examination
* Normal hematology values including hemoglobin, hematocrit, WBC, platelets, WBC differential
* Normal laboratory test including : Blood urea nitrogen, sGPT, sGOT, alkaline phosphatase, total bilirubin, total protein, fasting glucose, albumin and creatinine
* Normal urinalysis results including: specific gravity, color, pH, sugar, albumin, bilirubin, RBC, WBC and casts
* Acceptable electrocardiogram (ECG) result
* Negative result for serological tests of Hepatitis B, Hepatitis C and HIV
* Negative result for pregnancy test

Exclusion Criteria:

* Smoker or alcoholism
* Pregnant woman or nursing mother
* Have history of hepatic, cardiovascular, gastrointestinal or renal disease
* Potentially sensitive to azithromycin or other related drugs
* Received any investigation drug within four weeks
* Donation or loss more than 450 mL of blood within 3 months prior to the screening

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of azithromycin until 120 h after oral administration of 500 mg Azithromycin tablet (ng/mL) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Yahdiana Harahap, Prof, Principal Investigator — Indonesia University
Locations (1):
- PT Clinisindo Laboratories, Jakarta, Indonesia